CLINICAL TRIAL: NCT04190004
Title: Effect of Intranasal Vasopressin on Cooperative Behavior in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dr Naren P Rao, Additional Professor, National Institute of Mental Health and Neuro Sciences, India
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IEC/2017
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: After completion of clinical assessments all subjects will receive either 40 IU of vasopressin or saline in counterbalanced order on two separate days and perform the behavioral tasks
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vasopressin (Experimental): All subjects will receive bot 40IU of vasopressin and saline placebo in counterbalanced design
  Interventions: Drug: Vasopressins
- Placebo (Placebo Comparator): All subjects will receive bot 40IU of vasopressin and saline placebo in counterbalanced design
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vasopressins — 40 International units of vasopressin or placebo will be given intra-nasally. The order of the administration will be counterbalanced
  Arms: vasopressin
Drug: Placebo — 40 International units of vasopressin or placebo will be given intra-nasally. The order of the administration will be counterbalanced
  Arms: Placebo

SUMMARY:
The study investigates the effect of 40IU of intranasal vasopressin on cooperative behavior in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Diagnosed as Schizophrenia or Schizophreniform disorder as per DSM IV TR
* At least 7 years of formal education
* MOCA score >24

Exclusion Criteria:

* Diagnoses of SIADH, Diabetes Insipidus
* Substance dependence in the past 12 months, excluding nicotine dependence
* Current comorbid axis 1 psychiatric disorder
* Hypersensitivity or previous allergy to Vasopressin
* Serious medical or neurological illness which may interfere with assessment and administration of vasopressin
* Hypertension
* Impaired renal functions based on serum creatinine above 1.5
* Electrolyte imbalance
* Receiving ECT or has received ECT in the past 8 weeks
* Clinical history of mental retardation
* Pregnancy • Lactation
* Risk of harm to self or others
* Any significant nasal pathology which may hinder the intranasal absorption of the drug
* Hearing or visual impairment that significantly affects the comprehension and execution of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Performance in Dictator game | 60 minutes
  Amount of money shared in dictator game
Performance in stag hunt game | 60 minutes
  Security level in stag hunt game

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health and Neurosciecnes, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No